CLINICAL TRIAL: NCT02174627
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Roxadustat for the Treatment of Anemia in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: Safety and Efficacy Study of Roxadustat to Treat Anemia in Patients With Chronic Kidney Disease (CKD), Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5740C00001
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-11

CONDITIONS: Anemia
Keywords: Renal,; CKD,; Roxadustat,; anemia,; non-dialysis
MeSH Terms: conditions — Anemia | interventions — roxadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roxadustat (Experimental)
  Interventions: Drug: Roxadustat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxadustat — The initial study drug dose is 70 mg three times a week (TIW). The dose is subsequently adjusted to achieve and maintain Hb 11±1 g/dL.
  Arms: Roxadustat
Drug: Placebo — The initial study drug dose is 70 mg three times a week (TIW). The dose is subsequently adjusted to achieve and maintain Hb 11±1 g/dL.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of roxadustat for treatment of anemia in patients with chronic kidney disease not on dialysis

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study in anemic patients with Stage 3, 4 or 5 chronic kidney disease (CKD) who are not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Age ≥18 years at screening visit 1
3. eGFR <60 mL/min/1.73 m2, (calculated by central lab) corresponding to stage 3, 4 or 5CKD according to the Kidney Disease Outcomes Quality Initiative (KDOQI), not receiving dialysis
4. Mean of 2 most recent central laboratory Hb values during the screening period, obtained at least 7 days apart, must be <10.0 g/dL
5. Ferritin ≥50 ng/mL at randomization (obtained from screening visit)
6. TSAT ≥15 % at randomization (obtained from screening visit)
7. Serum folate level ≥ lower limit of normal (LLN) at randomization (obtained from screening visit)
8. Serum vitamin B12 level ≥LLN at randomization (obtained from screening visit)
9. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) and total bilirubin (Tbili) ≤1.5 x ULN at randomization (obtained from screening visit)
10. Body weight 45 to 160 kg

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous randomization in the present study
3. Any erythropoietin analogue treatment within 6 weeks of randomization
4. New York Heart Association Class III or IV congestive heart failure at enrollment
5. Myocardial infarction (MI), acute coronary syndrome, stroke, seizure or a thrombotic/thromboembolic event (e.g., deep vein thrombosis or pulmonary embolism) within 12 weeks prior to randomization
6. History of chronic liver disease (e.g., chronic infectious hepatitis, chronic auto- immune liver disease, cirrhosis or fibrosis of the liver)
7. Known hereditary hematologic disease such as thalassemia, sickle cell anemia, a history of pure red cell aplasia or other known causes for anemia other than CKD
8. Known and untreated retinal vein occlusion or known and untreated proliferative diabetic retinopathy (risk for retinal vein thrombosis)
9. Diagnosis or suspicion (e.g. complex kidney cyst of Bosniak Category IIF, III or IV) of renal cell carcinoma on renal ultrasound (or other imaging procedure e.g. CT scan or MRI) conducted at screening or within 12 weeks prior to randomization
10. Systolic BP ≥160 mmHg or diastolic BP ≥95 mmHg (confirmed by repeated measurement), within 2 weeks prior to randomization. Patients may be rescreened once BP controlled
11. History of prostate cancer, breast cancer or any other malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps
12. Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus antibody (anti-HCV Ab)
13. Chronic inflammatory diseases such as rheumatoid arthritis, systemic lupus erythematosus (SLE), ankylosing spondylitis, psoriatic arthritis or inflammatory bowel disease that is determined to be the principal cause of anemia
14. Known hemosiderosis, hemochromatosis or hypercoagulable condition
15. Any prior organ transplant or a scheduled organ transplantation date
16. Any red blood cell transfusion (RBC) during the screening period
17. Any current condition leading to active significant blood loss
18. Any treatment with roxadustat or a hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI)
19. Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within at least 1 month of the first administration of IP in this study. (Note: patients consented and screened, but not randomized in this study or a previous study are not excluded)
20. History of alcohol or drug abuse within 2 years prior to randomization
21. Females of childbearing potential, unless using contraception as detailed in the protocol or sexual abstinence
22. Pregnant or breastfeeding females
23. Known allergy to the investigational product or any of its ingredients
24. Any medical condition, including active, clinically significant infection, that in the opinion of the investigator or Sponsor may pose a safety risk to a patient in this study, which may confound efficacy or safety assessment or may interfere with study participation

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2781 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Fishbane, MD, Principal Investigator — Chief Division of Kidney Diseases and Hypertension, North Shore University Hospital, Great Neck, NY, USA; Mark Houser, MD, Study Director — AZ R&D Gaithersburg, USA
Locations (266):
- United States (75):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Bakersfield, California
  - Research Site, El Centro, California
  - Research Site, Escondido, California
  - Research Site, Glendale, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, National City, California
  - Research Site, Northridge, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Dimas, California
  - Research Site, San Francisco, California
  - Research Site, San Luis Obispo, California
  - Research Site, Upland, California
  - Research Site, Arvada, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Aventura, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Joliet, Illinois
  - Research Site, La Grange, Illinois
  - Research Site, Metairie, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Rockport, Maine
  - Research Site, Greenbelt, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Port Huron, Michigan
  - Research Site, Gulfport, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Rochester, New Hampshire
  - Research Site, Flushing, New York
  - Research Site, Great Neck, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Uniontown, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lufkin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, St. George, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Woodbridge, Virginia
- Argentina (13):
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, Ciudad Autónoma de Bs. As.
  - Research Site, Ciudadela
  - Research Site, La Plata
  - Research Site, Lanús
  - Research Site, Mar del Plata
  - Research Site, Munro
  - Research Site, Ramos Mejía
  - Research Site, Rosario
  - Research Site, San Isidro
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Rosa
- Brazil (10):
  - Research Site, Curitiba
  - Research Site, Feira de Santana
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Joinville
  - Research Site, Juiz de Fora
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
- Bulgaria (11):
  - Research Site, Botevgrad
  - Research Site, Dupnitsa
  - Research Site, Gotse Delchev
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Samokov
  - Research Site, Sandanski
  - Research Site, Silistra
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Yambol
- Canada (17):
  - Research Site, Edmonton, Alberta
  - Research Site, Kamloops, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, Sydney, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Whitby, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Colombia (4):
  - Research Site, Cali
  - Research Site, Chía
  - Research Site, Medellín
  - Research Site, Zipaquirá
- Czechia (10):
  - Research Site, Brno
  - Research Site, Havlíčkův Brod
  - Research Site, Ivančice
  - Research Site, Prague
  - Research Site, Rychnov nad Kněžnou
  - Research Site, Slaný
  - Research Site, Slavkov u Brna
  - Research Site, Šumperk
  - Research Site, Ústí nad Labem
  - Research Site, Ústí nad Orlicí
- Germany (3):
  - Research Site, Berlin
  - Research Site, Cloppenburg
  - Research Site, Cologne
- Hungary (12):
  - Research Site, Ajka
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Hatvan
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Polgár
  - Research Site, Salgótarján
  - Research Site, Siófok
  - Research Site, Tatabánya
  - Research Site, Velence
- India (15):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Chennai
  - Research Site, Ghaziabad NCR
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Maharashtra
  - Research Site, Mumbai
  - Research Site, Mysore
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Vijayawada
  - Research Site, Visakhapatnam
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Kubang Kerian
  - Research Site, Putrajaya
  - Research Site, Taiping
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Minatitlán
  - Research Site, Veracruz
  - Research Site, Xalapa
- Peru (4):
  - Research Site, Bellavista
  - Research Site, Ica
  - Research Site, Lima
  - Research Site, Trujillo
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Iloilo City
  - Research Site, Quezon City
- Poland (6):
  - Research Site, Ciechanów
  - Research Site, Gmina Końskie
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Sochaczew
  - Research Site, Tczew
- Puerto Rico (5):
  - Research Site, Cidra
  - Research Site, Rio Piedras
  - Research Site, Río Grande
  - Research Site, San Juan
  - Research Site, Toa Baja
- Romania (4):
  - Research Site, Arad
  - Research Site, Bucharest
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (13):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Perm
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Ufa
  - Research Site, Volgograd
- Slovakia (5):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Kráľovský Chlmec
  - Research Site, Nové Zámky
  - Research Site, Zvolen
- South Korea (9):
  - Research Site, Ansan-si
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
- Spain (5):
  - Research Site, Almería
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Khon Kaen
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (13):
  - Research Site, Chernivtsi
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Khmelnytsky
  - Research Site, Kirovograd
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Rivne
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
- Vietnam (5):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh
  - Research Site, Huế

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Provenzano R, Szczech L, Leong R, Saikali KG, Zhong M, Lee TT, Little DJ, Houser MT, Frison L, Houghton J, Neff TB. Efficacy and Cardiovascular Safety of Roxadustat for Treatment of Anemia in Patients with Non-Dialysis-Dependent CKD: Pooled Results of Three Randomized Clinical Trials. Clin J Am Soc Nephrol. 2021 Aug;16(8):1190-1200. doi: 10.2215/CJN.16191020. PMID 34362786
- [Derived] Fishbane S, El-Shahawy MA, Pecoits-Filho R, Van BP, Houser MT, Frison L, Little DJ, Guzman NJ, Pergola PE. Roxadustat for Treating Anemia in Patients with CKD Not on Dialysis: Results from a Randomized Phase 3 Study. J Am Soc Nephrol. 2021 Mar;32(3):737-755. doi: 10.1681/ASN.2020081150. Epub 2021 Feb 10. PMID 33568383
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5740C00001&attachmentIdentifier=e591fa4d-7259-4500-bf4c-783f4239fab9&fileName=D5740C00001_redacted_CSP_from_PRS.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5740C00001&attachmentIdentifier=cf047ffd-547d-4bee-b970-58c377627038&fileName=D5740C00001_SAP-v3_Redacted_28-Sep-2018.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 385 centers in 25 countries worldwide across the United States, Canada, Latin America, Asia and Europe between 26 June 2014 and 04 October 2018. Participants with chronic kidney disease who were not on dialysis were recruited in this study.
Pre-assignment Details: Study had a screening period (up to 6 weeks), treatment period (up to 4 years) and follow-up period (4 weeks after treatment period for those who completed treatment). 2781 participants were randomized, of which 2761 were included in the analysis and 20 were excluded. Only participants included in the analysis are presented in the participant flow.
Groups:
- Roxadustat: Participants received roxadustat tablets orally three times a week (TIW). The initial dose was 70 milligram (mg) TIW and was titrated to achieve and maintain haemoglobin (Hb) 11±1 grams per deciliter (g/dL). Treatment started on Day 1 and treatment duration was variable for individual participants (estimated up to 4 years). Dose adjustments were permitted starting at Week 4 and at intervals of every 4 weeks until Week 52, every 8 weeks thereafter using a dose adjustment algorithm; all dose adjustments were based on Hb values.
- Placebo: Participants received placebo tablets orally TIW. Dosing instructions were matched to instructions provided for roxadustat (ie, initial dose matched to 70 mg TIW). Treatment started on Day 1 and treatment duration was variable for individual participants (estimated up to 4 years). Dose adjustments were permitted starting at Week 4 and at intervals of every 4 weeks until Week 52, every 8 weeks thereafter using a dose adjustment algorithm; all dose adjustments were based on Hb values.
Period: Overall Study
Arm/Group | Roxadustat | Placebo
Started (Randomized and included in the analysis) | 1384 | 1377
Received Treatment | 1384 | 1376
Discontinued Treatment | 499 | 801
Completed (Completed the study) | 1300 | 1247
Not Completed | 84 | 130
Not completed — Missing | 0 | 1
Not completed — Incorrect enrolment before randomization | 0 | 1
Not completed — Participant decision | 84 | 128

BASELINE CHARACTERISTICS:
Population: The Intention-To-Treat (ITT) analysis set included all participants who were randomized to investigational product (IP) irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis.
Groups:
- Roxadustat: Participants received roxadustat tablets orally TIW. The initial dose was 70 mg TIW and was titrated to achieve and maintain Hb 11±1 g/dL. Treatment started on Day 1 and treatment duration was variable for individual participants (estimated up to 4 years). Dose adjustments were permitted starting at Week 4 and at intervals of every 4 weeks until Week 52, every 8 weeks thereafter using a dose adjustment algorithm; all dose adjustments were based on Hb values.
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Placebo | Total
Number analyzed (Participants) | 1384 | 1377 | 2761
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (14.67) | 62.4 (14.14) | 61.7 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 820 | 774 | 1594
  Male | 564 | 603 | 1167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 344 | 357 | 701
  Not Hispanic or Latino | 1040 | 1020 | 2060
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 623 | 611 | 1234
  Black or African American | 112 | 115 | 227
  Asian | 544 | 538 | 1082
  Native Hawaiian or other Pacific Islander | 0 | 2 | 2
  American Indian or Alaska Native | 24 | 29 | 53
  Other | 81 | 82 | 163

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hb Averaged Over Week 28 to Week 52
Description: Baseline Hb was defined as the mean of the last 3 central laboratory Hb values from the screening and randomization visits. Mean change in Hb from baseline to mean value from Week 28 to Week 52 was analyzed using a missing at random (MAR) based multiple imputation analysis of covariance (ANCOVA) model with baseline Hb, baseline estimated glomerular filtration rate (eGFR), cardiovascular (CV) history, geographic region and treatment group as fixed effect covariates. The adjusted least squares (LS) mean estimates of change from baseline to mean during Week 28 to Week 52 are presented.
Time Frame: Baseline (Day 1, Week 0) and Week 28 to Week 52.
Population: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1334 | 1330
g/dL | 1.75 (0.033) | 0.40 (0.034)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; MAR-based multiple imputation ANCOVA model; Test type: Superiority — Superiority of roxadustat compared with placebo would be declared if the lower bound of the 2-sided 95% confidence interval (CI) of the difference between roxadustat and placebo exceeded 0 g/dL; p < 0.001, ANCOVA; LS Mean Difference = 1.35, 95% CI 2-sided [1.27 to 1.43], Standard Error of Mean 0.041

2. Secondary Outcome: Percentage of Participants With Hb Response During the First 24 Weeks of Treatment
Description: Hb response was defined as:
  * Hb ≥ 11.0 g/dL and Hb increase from baseline by ≥ 1.0 g/dL for participants with baseline Hb > 8.0 g/dL; or
  * Hb increase from baseline by ≥ 2.0 g/dL, for participants with baseline Hb ≤ 8.0 g/dL at 2 consecutive visits (with available data) separated at least 5 days during the first 24 weeks of treatment without having received rescue therapy (red blood cell [RBC] transfusion, erythropoietin analogue, or intravenous [IV] iron) prior to Hb response. The percentage of participants with an Hb response during the first 24 weeks of treatment is presented.
Time Frame: Baseline (Day 1, Week 0) up to Week 24.
Population: The Full Analysis Set (FAS) included all participants in the ITT analysis set who received at least 1 dose of IP and had baseline Hb and at least 1 post-dose Hb assessment. Participants from the FAS, with data available for analysis are presented.
Measure: Number; unit: Percentage of participants
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1371 | 1357
Percentage of participants | 77.0 | 8.5
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Comparison of the percentage of responders for roxadustat versus placebo was analysed using a Cochran-Mantel-Haenszel test adjusting for baseline Hb, baseline eGFR, geographic region and CV history; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Relative Risk = 9.12, 95% CI 2-sided [7.63 to 10.89]

3. Secondary Outcome: Mean Change From Baseline in Hb Averaged Over Week 28 to Week 52 in Participants With Baseline High Sensitivity C-Reactive Protein (hsCRP) Greater Than the Upper Limit of Normal (ULN)
Description: Baseline hsCRP was quantified from stored biomarker samples obtained at randomization. Baseline Hb was defined as the mean of the last 3 central laboratory Hb values from the screening and randomization visits. Mean change in Hb from baseline to mean value during Week 28 to Week 52 was analyzed using a MAR based multiple imputation ANCOVA model with baseline Hb, baseline eGFR, CV history, geographic region and treatment group as fixed effect covariates. The adjusted LS mean estimates of change from baseline in participants with baseline hsCRP >ULN to mean during Week 28 to Week 52 are presented.
Time Frame: Baseline (Day 1, Week 0) and Week 28 to Week 52.
Population: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis. Only participants who consented to the use of donated biomarker samples and had baseline hsCRP >ULN were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 213 | 198
g/dL | 1.75 (0.087) | 0.62 (0.091)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; MAR-based multiple imputation ANCOVA model; Test type: Superiority — Superiority of roxadustat compared with placebo would be declared if the lower bound of the 2-sided 95% CI of the difference between roxadustat and placebo exceeded 0 g/dL; p < 0.001, ANCOVA; LS Mean Difference = 1.13, 95% CI 2-sided [0.91 to 1.35], Standard Error of Mean 0.112

4. Secondary Outcome: Proportion of Total Time of Interpolated Hb Values Greater Than or Equal To 10 g/dL From Week 28 to Week 52
Description: Proportion of total time of interpolated Hb values ≥10 g/dL was calculated as the time the linearly interpolated curve between measurements ≥10 g/dL divided by the time between measurements from Week 28 to Week 52. Proportion of total time was analyzed using an ANCOVA model with baseline Hb and baseline eGFR as covariates, and CV history, geographic region and treatment group as fixed effects. The adjusted LS mean estimates of change from Week 28 to Week 52 are presented.
Time Frame: Week 28 up to Week 52.
Population: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis. Participants without any Hb measurements from Week 28 were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: proportion of total time
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1220 | 1145
proportion of total time | 0.82 (0.011) | 0.33 (0.011)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; ANCOVA model; Test type: Superiority — Superiority of roxadustat compared with placebo would be declared if the lower bound of the 2-sided 95% CI of the difference between roxadustat and placebo exceeded 0; p < 0.001, ANCOVA; LS Mean Difference = 0.50, 95% CI 2-sided [0.47 to 0.52], Standard Error of Mean 0.013

5. Secondary Outcome: Proportion of Total Time of Interpolated Hb Values Within the Interval of 10 to 12 g/dL From Week 28 to Week 52
Description: Proportion of total time of interpolated Hb values within the interval of 10 to 12 g/dL was calculated as the time the linearly interpolated curve between measurements were within 10 to 12 g/dL divided by the time between measurements from Week 28 to Week 52. Proportion of total time was analyzed using an ANCOVA model with baseline Hb and baseline eGFR as covariates, and CV history, geographic region and treatment group as fixed effects. The adjusted LS mean estimates of change from Week 28 to Week 52 are presented.
Time Frame: Week 28 up to Week 52.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: proportion of total time
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1220 | 1145
proportion of total time | 0.70 (0.010) | 0.28 (0.010)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; ANCOVA model; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = 0.42, 95% CI 2-sided [0.40 to 0.45], Standard Error of Mean 0.013

6. Secondary Outcome: Mean Change in Low-Density Lipoprotein (LDL) Cholesterol From Baseline to Week 24
Description: Baseline LDL was defined as the last result obtained prior to randomization. Mean changes in LDL cholesterol from baseline to Week 24 was analyzed using an ANCOVA model with baseline LDL, baseline Hb and baseline eGFR as covariates, and CV history, geographic region and treatment group as fixed effects. The adjusted LS mean estimates of change from baseline to Week 24 are presented.
Time Frame: Baseline (Day 1, Week 0) and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimole per liter
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1147 | 1133
millimole per liter | -0.38 (0.028) | -0.02 (0.027)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; ANCOVA model; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p < 0.001, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.42 to -0.29], Standard Error of Mean 0.033

7. Secondary Outcome: Time-To-First Instance of Receiving IV Iron, RBC Transfusion or Erythropoietin Analogue as Rescue Therapy
Description: Time-to-first rescue therapy (IV iron, RBC transfusion or erythropoietin analogue) was calculated as (date of first rescue therapy, or date of censoring if no rescue therapy was taken) minus (date of first dose of IP) +1. Event rate was calculated as (number of participants with event) divided by (the total number of days at risk for event across all participants in given group divided by 365.25) multiplied by 100. The event rate is presented for participants with events.
Time Frame: Baseline (Day1, Week 0) up to End of Study (EOS) visit (4 weeks after the treatment period) (or up to date of first rescue therapy), with treatment duration up to 4 years.
Population: The on-treatment plus 28 days (OT+28) analysis set included all participants who received at least 1 dose of randomized IP, except for those excluded from analysis. Participants were censored 28 days after last intake of IP.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1384 | 1376
Events per 100 participant years | 11.90 | 39.76
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Treatments were compared using a Cox proportional hazards model, with baseline Hb and baseline eGFR as continuous variables used as covariates, and treatment group, CV history and geographic region as fixed effects. The Efron method was used for ties and p-values were calculated using the Wald test; Test type: Superiority — Superiority of roxadustat compared with placebo would be declared if the upper limit of the 2-sided 95% CI for the HR was ≤1.0; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.26, 95% CI 2-sided [0.23 to 0.31]

8. Secondary Outcome: Time-To-First Instance of Receiving a RBC Transfusion As Rescue Therapy
Description: Time-to-first RBC rescue therapy was calculated as (date of first RBC rescue therapy, or date of censoring if no rescue therapy was taken) minus (date of first dose of IP) +1. Event rate was calculated as (number of participants with event) divided by (the total number of days at risk for event across all participants in given group divided by 365.25) multiplied by 100. The event rate is presented for participants with events.
Time Frame: Baseline (Day1, Week 0) up to EOS visit (4 weeks after the treatment period) (or up to date of first RBC rescue therapy), with treatment duration up to 4 years.
Population: The OT+28 analysis set included all participants who received at least 1 dose of randomized IP, except for those excluded from analysis. Participants were censored 28 days after last intake of IP.
Measure: Number; unit: Events per 100 participant years
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1384 | 1376
Events per 100 participant years | 7.98 | 19.61
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.30 to 0.44]

9. Secondary Outcome: Mean Change From Baseline in Short Form 36 (SF-36) Vitality Sub-Score From Week 12 to Week 28
Description: SF-36 is a Quality of Life (QoL) scale comprising 8 domains of health status: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health. Each domain score is on a scale from 0-100 (worst health possible to best health possible); higher scores indicate better health status. Mean change in SF-36 Vitality sub-score from baseline to mean from Week 12 to Week 28 was analyzed using a mixed model for repeated measures (MMRM) with terms for baseline score, treatment group, baseline Hb, baseline eGFR, CV history, geographic region, visit and treatment-by-visit interaction as fixed effects and participant as random effect. The adjusted LS mean estimates of change from baseline to mean score from Week 12 to Week 28 are presented.
Time Frame: Baseline (Day 1, Week 0) and Week 12 to Week 28.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1279 | 1235
scores on a scale | 1.59 (0.231) | 1.15 (0.233)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; MMRM analysis; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.120, Mixed Models Analysis; LS Mean Difference = 0.44, 95% CI 2-sided [-0.11 to 0.99], Standard Error of Mean 0.283

10. Secondary Outcome: Annual Rate of eGFR Change From Baseline Prior to the Initiation of Dialysis or Kidney Transplant
Description: Baseline eGFR was defined as the mean of all available central laboratory values prior to or at randomization. Rate of change in eGFR from baseline during the entire treatment period (in millilitres/minute/1.73 meters squared/years [mL/min/1.73m^2/years]) was estimated using a random effects model using all post-baseline eGFR values prior to initiation of dialysis/transplant. Baseline eGFR, baseline Hb, geographic region, CV history, treatment group and post-baseline eGFR measurement time were used as fixed effects and participant and time (years) as random effects, ie, random intercept and slope.
Time Frame: Baseline (Day1, Week 0) up to EOS visit (4 weeks after the treatment period), with treatment duration up to 4 years.
Population: as for outcome 1
Measure: Number; unit: eGFR rate (mL/min/1.73m^2/years)
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1326 | 1314
eGFR rate (mL/min/1.73m^2/years) | -3.70 | -3.19
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in rate of change in eGFR; random effects analysis; Test type: Other; p = 0.046, Random Effects Analysis — Nominal p-value (as prior sequential outcome measure p-value did not meet < 0.05; Rate of Change Difference = -0.51, 95% CI 2-sided [-1.00 to -0.01], Standard Error of Mean 0.254

11. Secondary Outcome: Mean Change From Baseline in SF-36 Physical Functioning Sub-Score From Week 12 to Week 28
Description: SF-36 is a QoL scale comprising 8 domains of health status: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional and Mental Health. Each domain score is on a scale from 0-100 (worst health possible to best health possible); higher scores indicate better health status. Mean change in SF-36 Physical Functioning sub-score from baseline to mean from Week 12 to Week 28 was analyzed using a MMRM with terms for baseline score, treatment group, baseline Hb, baseline eGFR, CV history, geographic region, visit and treatment-by-visit interaction as fixed effects and participant as random effect. The adjusted LS mean estimates of change from baseline to mean score from Week 12 to Week 28 are presented.
Time Frame: Baseline (Day 1, Week 0) and Week 12 to Week 28.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Roxadustat | Placebo
Number analyzed (Participants) | 1279 | 1234
scores on a scale | 0.14 (0.222) | -0.39 (0.224)
Statistical Analysis 1: Comparison: Roxadustat vs Placebo; Difference between groups (roxadustat minus placebo) in LS mean changes; MMRM analysis; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.051, Mixed Models Analysis — Nominal p-value (as prior sequential outcome measure p-value did not meet < 0.05; LS Mean Difference = 0.52, 95% CI 2-sided [0.00 to 1.05], Standard Error of Mean 0.269

ADVERSE EVENTS:
Time Frame: From date of randomization up to EOS visit (4 weeks after the treatment period), with treatment duration up to 4 years.
Description: The ITT analysis set included all participants who were randomized to IP irrespective of their protocol adherence and continued participation in the study, except for those excluded from analysis. All-Cause Mortality represents all deaths due to any cause.
Arm/Group | Roxadustat | Placebo
All-Cause Mortality (participants affected / at risk) | 284/1384 | 245/1377
Serious Adverse Events (participants affected / at risk) | 795/1384 | 749/1377
Other Adverse Events (participants affected / at risk) | 839/1384 | 757/1377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=1384) | Placebo (N=1377)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Evans syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypocoagulable state (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 8 (8) | 5 (5)
Acute left ventricular failure (Cardiac disorders) | 5 (6) | 4 (4)
Acute myocardial infarction (Cardiac disorders) | 26 (28) | 27 (31)
Angina pectoris (Cardiac disorders) | 10 (10) | 9 (9)
Angina unstable (Cardiac disorders) | 10 (10) | 10 (11)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 6 (6) | 3 (3)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 10 (10) | 12 (15)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 3 (4)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 9 (9) | 4 (4)
Cardiac asthma (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 25 (31) | 32 (35)
Cardiac failure acute (Cardiac disorders) | 8 (8) | 14 (16)
Cardiac failure chronic (Cardiac disorders) | 4 (4) | 5 (6)
Cardiac failure congestive (Cardiac disorders) | 33 (41) | 31 (42)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 6 (6) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 12 (12) | 7 (7)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Heart valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Metabolic cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 14 (14) | 13 (13)
Myocardial ischaemia (Cardiac disorders) | 4 (4) | 8 (8)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 2 (2)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 2 (3)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vestibular ataxia (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 5 (5) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 3 (3) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 2 (2)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 2 (2)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 5 (5)
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 4 (5) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 18 (24) | 15 (18)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 20 (20) | 15 (16)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhagic ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (2) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 4 (5) | 3 (4)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 5 (5)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (2) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 5 (5) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4) | 4 (4)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal cloudy effluent (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (11) | 4 (4)
Uraemic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Asthenia (General disorders) | 13 (14) | 9 (9)
Catheter site haemorrhage (General disorders) | 0 (0) | 2 (2)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 43 (43) | 28 (28)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2)
Generalised oedema (General disorders) | 17 (25) | 7 (11)
Hernia pain (General disorders) | 0 (0) | 1 (1)
Implant site extravasation (General disorders) | 1 (1) | 0 (0)
Implant site necrosis (General disorders) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2)
Oedema (General disorders) | 7 (9) | 7 (7)
Oedema due to renal disease (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 7 (10) | 5 (10)
Pacemaker generated arrhythmia (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 5 (5)
Stenosis (General disorders) | 0 (0) | 1 (2)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 5 (5) | 11 (11)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 4 (6) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 2 (2)
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Device allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 2 (3) | 1 (1)
Renal transplant failure (Immune system disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 3 (3) | 3 (3)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 5 (5)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 3 (3) | 3 (3)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 2 (2)
Arthritis bacterial (Infections and infestations) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 4 (4) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bone tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 7 (7) | 9 (9)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cardiac valve abscess (Infections and infestations) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 3 (3) | 8 (9)
Cellulitis (Infections and infestations) | 24 (27) | 13 (13)
Cellulitis gangrenous (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 4 (4) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus nephritis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 14 (14) | 5 (6)
Device related sepsis (Infections and infestations) | 3 (4) | 5 (5)
Diabetic foot infection (Infections and infestations) | 1 (1) | 4 (4)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (3)
Diarrhoea infectious (Infections and infestations) | 4 (4) | 4 (5)
Diverticulitis (Infections and infestations) | 4 (7) | 3 (3)
Emphysematous cystitis (Infections and infestations) | 1 (1) | 1 (2)
Emphysematous pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Endotoxic shock (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 10 (10) | 7 (9)
Gastroenteritis (Infections and infestations) | 13 (16) | 8 (8)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 2 (2) | 2 (2)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected lymphocele (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 5 (5)
Intestinal tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 2 (4) | 5 (5)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Lung abscess (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 3 (3) | 2 (3)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 1 (2) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Parvovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Perinephric abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 15 (17) | 14 (19)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pleural infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 113 (149) | 88 (107)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 3 (3)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 2 (2)
Purulence (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 8 (9) | 5 (5)
Pyelonephritis acute (Infections and infestations) | 6 (6) | 4 (4)
Pyelonephritis chronic (Infections and infestations) | 11 (14) | 11 (14)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 3 (5) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 49 (51) | 23 (24)
Septic shock (Infections and infestations) | 18 (19) | 15 (15)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 3 (3)
Stenotrophomonas sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 4 (4)
Taeniasis (Infections and infestations) | 1 (4) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (2) | 0 (0)
Tuberculosis (Infections and infestations) | 5 (5) | 3 (4)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 36 (38) | 26 (32)
Urinary tract infection bacterial (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 8 (11) | 6 (6)
Vascular access site infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 3 (3)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 18 (19) | 9 (9)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dialysis disequilibrium syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dialysis related complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spleen contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 6 (7) | 2 (2)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anticoagulation drug level increased (Investigations) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Blood urine present (Investigations) | 1 (2) | 0 (0)
Coagulation factor decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Calciphylaxis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 6 (10) | 10 (12)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 20 (28) | 22 (27)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Food aversion (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 16 (17) | 9 (10)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 41 (53) | 25 (35)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 32 (38) | 26 (27)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (8) | 6 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 9 (9) | 3 (3)
Cerebral infarction (Nervous system disorders) | 13 (14) | 8 (9)
Cerebrovascular accident (Nervous system disorders) | 15 (15) | 11 (11)
Cerebrovascular disorder (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cervical cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 2 (2)
Coma uraemic (Nervous system disorders) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2) | 0 (0)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic hyperosmolar coma (Nervous system disorders) | 1 (1) | 1 (1)
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (2)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (5) | 2 (2)
Encephalopathy (Nervous system disorders) | 5 (5) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Facial spasm (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 9 (9) | 7 (7)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Lacunar stroke (Nervous system disorders) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraparesis (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post stroke seizure (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 6 (6) | 2 (3)
Senile dementia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 3 (3)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 5 (5)
Uraemic encephalopathy (Nervous system disorders) | 2 (2) | 2 (2)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Vestibular migraine (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (2)
Device failure (Product Issues) | 2 (3) | 0 (0)
Device malfunction (Product Issues) | 3 (4) | 2 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 3 (4) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Vascular cognitive impairment (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 41 (48) | 32 (33)
Anuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 61 (73) | 60 (79)
Chronic kidney disease (Renal and urinary disorders) | 8 (8) | 7 (7)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (2) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 199 (211) | 201 (211)
Glomerulonephritis (Renal and urinary disorders) | 1 (2) | 1 (1)
Glomerulonephritis chronic (Renal and urinary disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephritic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 1 (1)
Oedematous kidney (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal atrophy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 3 (4)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 4 (5) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal papillary necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal pelvis fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 2 (2)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (3)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 5 (5) | 1 (1)
Urinary tract inflammation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatic mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 22 (25)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 20 (20)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 3 (3)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 16 (20)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 16 (16)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (9)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (6)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic rupture (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (2) | 4 (4)
Arteriosclerosis (Vascular disorders) | 2 (2) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 15 (15) | 4 (4)
Distributive shock (Vascular disorders) | 1 (1) | 1 (1)
Dry gangrene (Vascular disorders) | 0 (0) | 2 (2)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (2) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 4 (4)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 17 (19) | 16 (16)
Hypertensive crisis (Vascular disorders) | 33 (51) | 27 (31)
Hypertensive emergency (Vascular disorders) | 21 (24) | 21 (23)
Hypotension (Vascular disorders) | 6 (6) | 8 (8)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 6 (6)
Iliac artery perforation (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Paget-Schroetter syndrome (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 5 (5) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (2) | 3 (4)
Peripheral artery stenosis (Vascular disorders) | 2 (2) | 1 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 4 (6) | 2 (4)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 4 (4)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Visceral congestion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=1384) | Placebo (N=1377)
Constipation (Gastrointestinal disorders) | 91 (126) | 88 (101)
Diarrhoea (Gastrointestinal disorders) | 138 (190) | 117 (156)
Nausea (Gastrointestinal disorders) | 124 (171) | 103 (127)
Vomiting (Gastrointestinal disorders) | 75 (90) | 67 (85)
Oedema peripheral (General disorders) | 144 (192) | 106 (135)
Bronchitis (Infections and infestations) | 72 (80) | 64 (76)
Upper respiratory tract infection (Infections and infestations) | 95 (137) | 75 (100)
Urinary tract infection (Infections and infestations) | 152 (205) | 94 (135)
Viral upper respiratory tract infection (Infections and infestations) | 101 (159) | 106 (152)
Hyperkalaemia (Metabolism and nutrition disorders) | 86 (105) | 75 (86)
Arthralgia (Musculoskeletal and connective tissue disorders) | 73 (85) | 53 (61)
Back pain (Musculoskeletal and connective tissue disorders) | 70 (87) | 57 (69)
Dizziness (Nervous system disorders) | 74 (91) | 86 (113)
Headache (Nervous system disorders) | 93 (122) | 82 (96)
End stage renal disease (Renal and urinary disorders) | 93 (93) | 87 (88)
Cough (Respiratory, thoracic and mediastinal disorders) | 105 (123) | 69 (91)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 70 (85) | 64 (80)
Pruritus (Skin and subcutaneous tissue disorders) | 68 (84) | 80 (89)
Hypertension (Vascular disorders) | 148 (190) | 117 (151)

LIMITATIONS AND CAVEATS:
20 participants were excluded from the analysis due to Good Clinical Practice violations or system technical issues (9 in roxadustat group and 11 in placebo group). Higher IP discontinuation was observed in placebo group versus in roxadustat group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT02174627/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT02174627/SAP_001.pdf